CLINICAL TRIAL: NCT04164108
Title: Pilot Study to Assess the Feasibility and Safety of Intermittent Enteral Feeding in Mechanically Ventilated Medical Intensive Care Unit Patients
Brief Title: Pilot: Feasibility of Intermittent Enteral Feeding in Ventilated MICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB Exempt
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Nutrition
Keywords: intensive care unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent feed participants (Experimental): Patients admitted to medical ICU #1 (of 2 at our hospital) will be assigned to receive intermittent enteral feeding protocol. They will receive four equal volume feeds at 8:00, 12:00, 16:00, and 20:00 hours.
  Interventions: Dietary Supplement: Intermittent Enteral Nutrition Protocol
- Control participants (No Intervention): Patients admitted to the medical ICU #2 (of 2 at our hospital) will receive usual care.

INTERVENTIONS:
Dietary Supplement: Intermittent Enteral Nutrition Protocol — Patients will receive total recommended nutrition divided into four equal meals, delivered at a rate of 400 cc/hr at 8:00, 12:00, 16:00, 20:00. Titration schedule will include administering 50% of volume for first two feeds, then 75%, and then 100%.
  Arms: Intermittent feed participants

SUMMARY:
Specific Aims:

Aim 1: Evaluate the feasibility of intermittent feeding in intensive care unit patients who are mechanically ventilated.

Aim 2: Evaluate the safety and patient tolerance of intermittent feeding in intensive care unit patients who are mechanically ventilated.

Aim 3: Determine efficacy of intermittent feeding in provision of required nutrition in mechanically ventilated intensive care unit patients.

Aim 4: Determine association of intermittent enteral feeding with glycemic control in mechanically ventilated intensive care unit patients.

DETAILED DESCRIPTION:
With the advent of the feeding pump, default enteral nutrition schedules in many medical intensive care units has shifted from intermittent or bolus feeding to continuous feeds. Clinical studies suggest that each of these strategies of providing nutrition is safe for patients with no significant difference in glycemic control or adverse effects. There is also data to suggest that approximating a more physiologic nutrition schedule with periods of feeding and periods of fasting may optimize gastrointestinal and metabolic hormonal feedback loops thereby effecting outcomes such as gastrointestinal motility, protein synthesis, and glycemic control, among others. Circadian rhythm research supports a temporally restricted period of feeding as well. Furthermore, periods of scheduled fasting will allow for provision of care that is incompatible with enteral feeds, without interrupting administration of nutrition (for example, procedures or testing, incompatible medications, etc).

Aims 1 and 2 will clarify whether an intermittent enteral nutrition schedule is acceptable to ICU staff and patients. Aims 3 and 4 will test whether this enteral feeding schedule is effective in providing patients with required nutrition and acceptable glycemic control.

This pilot will set the stage for a randomized controlled trial further investigating superiority of intermittent feeding as compared with the current standard of continuous feeding.

ELIGIBILITY:
Inclusion Criteria:

* Medical intensive care unit patients located in Yale-New Haven Hospital, York Street campus, North Pavilion 9 or 10.
* Hospitalized for less than or equal to 72 hours.
* Patients who are mechanically ventilated via endotracheal tube for at least 24 hours.
* Patients must have enteral access (nasogastric tube, orogastric tube).
* Team plans to initiate tube feeds.

Exclusion Criteria:

* Prior upper gastrointestinal surgery (including but not limited to gastric bypass surgery, gastric banding, complete or partial gastrectomy, Whipple procedure; cholecystectomy is acceptable).
* Chronic enteral nutrition (prior to current admission).
* History of significant esophageal dysmotility (history of GERD is acceptable).
* Unable to have head of bed elevated at least 30 degrees while intubated and being fed (this is standard protocol).
* Enteral access terminates post-pyloric (ie nasojejunal or jejunostomy tubes are to be excluded).
* Pre-existing percutaneous gastrostomy tube.
* History of small bowel obstruction or ileus on current admission.
* History of gastroparesis.
* Clinical care team is not planning to initiate enteral nutrition.
* At risk of refeeding syndrome.
* Pregnant patients.
* Patients receiving neuromuscular blockade.
* Patients with glycemic emergency (HHNK, DKA, severe hypoglycemia resulting in MICU admission).
* Patients otherwise excluded by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Proportion complete protocol | Up to 7 days
  This is defined as the proportion of patients who continue to receive intermittent enteral feeds during the entire course of their enteral nutrition or seven days, whichever comes first.

SECONDARY OUTCOMES:
Proportion correct pump rate | Up to 7 days
  This is defined as the proportion of the feeds that enteral feeding pump provides nutrition at appropriate rate.
Proportion clogged enteral access | Up to 7 days
  This is defined as the proportion of patients whose enteral access is clogged.
Proportion completed meals | Up to 7 days
  This is defined as the proportion of meals that are delivered.
Staff satisfaction | Up to 7 days
  This will be measured using a qualitative survey of bedside nurses and ICU nutritionists regarding perceptions of intervention feasibility.
Proportion held to accommodate a medication | Up to 7 days
  This is defined as the proportion of patients who had enteral nutrition held to accommodate a medication.
Proportion held to accommodate a procedure | Up to 7 days
  This is defined as the proportion of patients who had enteral nutrition held to accommodate a procedure.
Early mobility | Up to 7 days
  This is defined as the proportion of patients able to participate in early mobility.
Proportion feeding intolerance | Up to 7 days
  This is defined as the proportion of patients with one or more of the following conditions:
  * New onset nausea or vomiting
  * Clinical concern for ileus or obstruction, as documented in progress notes
  * New onset abdominal distension, as documented in progress notes
  * Abdominal X-ray (not obtained for purposes of line/tube placement verification)
Proportion Diarrhea | Up to 7 days
  This is defined as the proportion of patients with diarrhea.
Symptomatic elevated gastric residual volume | Up to 7 days
  This is defined as the proportion of patients with gastric residual volume >500 AND any of the following symptoms:
  * New onset nausea or vomiting
  * Clinical concern for ileus or obstruction, as documented in progress notes
  * New onset abdominal distension, as documented in progress notes
  * Abdominal X-ray (not obtained for purposes of line/tube placement verification)
Percent of recommended nutrition delivered | Up to 7 days
  This is defined as the average daily calorie intake as percentage of goal calories (determined by RD).
Nutrition delay | Up to 7 days
  This is defined as the time (hours) from intubation to patient receiving 50% of caloric needs.
Adequate nutrition provision | Up to 7 days
  This is defined as the proportion of days that patient is receiving enteral nutrition that at least 70% of caloric need is administered.
Inadequate nutrition provision | Up to 7 days
  This is defined as the proportion of days that patient is receiving enteral nutrition that less than 30% of caloric need is administered.
Hyperglycemia proportion | Up to 7 days
  This is defined as the proportion of glucose measurements closest to 8:00, 12:00, 16:00, 20:00 (including on basic metabolic panel and point of care testing) that are greater than or equal to 180.
Insulin drip usage | Up to 7 days
  This is defined as the proportion of glucose measurements closest to 8:00, 12:00, 16:00, 20:00 (including on basic metabolic panel and point of care testing) that are less than or equal to 60.
Non-diabetic insulin usage proportion | Up to 7 days
  This is defined as the proportion of patients who do not have a pre-existing diagnosis of diabetes mellitus who require any insulin dose.

CONTACTS AND LOCATIONS:
Overall Officials: Shyoko Honiden, MD, Principal Investigator — Program Director, Pulmonary & Critical Care Medicine Program, Internal Medicine
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale New Haven Hospital, York Street Campus, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No